CLINICAL TRIAL: NCT02392364
Title: Treat and Extend Versus Dosing Every Eight Weeks With Intravitreal Aflibercept Injections for the Treatment of Diabetic Macular Edema (EVADE Study)
Brief Title: Variable Interval Versus Set Interval Aflibercept for DME
Acronym: EVADE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-01-CRC
Record Dates: First submitted 2015-03-02; First posted 2015-03-19 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Cystoid Macular Edema; Diabetic Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Variable Treatment Dosing Arm (Active Comparator): Group 1 will receive injections every 4 weeks until diabetic macular edema on the OCT is decreased and stable. At that point, the length of time between injections may increase, depending on how the study eye is doing. The interval between study eye treatments may maintain, increase, or decrease once the variable treatment dosing has begun. This will be determined by an algorithm designed into a computer program
  Interventions: Drug: Intravitreal Aflibercept Injection
- Monthly Treatment Arm (Active Comparator): Group 2 will receive 5 intravitreal injections, monthly, for the first 5 months of the study. After those initial injections, visits/treatment will be every 8 weeks.
  Interventions: Drug: Intravitreal Aflibercept Injection

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection

SUMMARY:
The purpose of this study is to compare the safety and efficacy of intravitreal Eylea injections at a set interval, versus a variable dosing schedule (likely longer than one month), based on a specific individual's disease progression. There will be approximately 50 men and women at least 18 years of age, diagnosed with type 1 or type 2 diabetes, taking part in this study at 5 locations in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years and older with Type 1 or Type 2 diabetes mellitus
2. Patients with diabetic macular edema involving the center of the macular in the study eye (CST must measure at least 350µm on Heidelberg SDOCT, or 333µm on Cirrus SDOCT)
3. Decrease in vision determined to be primarily due to DME in the study eye
4. BCVA ETDRS letter score 78 to 24 (20/32 to 20/320) in the study eye
5. Willing and able to comply with clinical visits and study related procedures
6. Willing and able to provide signed informed consent

Exclusion Criteria:

1. History of vitreoretinal surgery in the study eye
2. Laser photocoagulation (panretinal or macular) in the study eye within 90 days of baseline
3. Previous use of intraocular or periocular corticosteroids in the study eye within 90 days of baseline
4. History of intravitreal anti-VEGF treatments in the study within 90days prior to baseline (not including prior intravitreal aflibercept injection [see exclusion criteria #5])
5. Any history of intravitreal aflibercept
6. Active proliferative diabetic retinopathy (PDR) in the study eye
7. History of idiopathic or autoimmune uveitis in the study eye
8. Cataract surgery in the study eye within 90 days of baseline
9. Aphakia in the study eye
10. Yttrium aluminum garnet (YAG) capsulotomy in the study eye within 30 days of baseline
11. Any intraocular surgery in the study eye within 90 days of day 1
12. Vitreomacular traction or epiretinal membrane in the study eye that is thought to affect central vision
13. Current iris neovascularization, vitreous hemorrhage, or traction retinal detachment in the study eye
14. Pre-retinal fibrosis involving the macula in the study eye
15. Uncontrolled glaucoma (defined as any patient who has had filtration surgery in the past, or likely to need filtration surgery in the future, or has IOP ≥30mmHg)
16. Myopia of a spherical equivalent prior to any possible refractive or cataract surgery of ≥-8 diopters
17. Concurrent disease in the study eye, other than DME, that could compromise BCVA, require medical or surgical intervention during the study period, or could confound interpretation of the results (including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause)
18. Ocular media of insufficient quality to obtain fundus and SDOCT images
19. Current treatment for a systemic infection
20. Administration of systemic anti-angiogenic agents within 180 days of baseline
21. Uncontrolled diabetes mellitus, in the opinion of the investigator
22. Uncontrolled blood pressure (define as systolic >180mmHg, or diastolic >110mmHg while patient is sitting)
23. History of CVA or MI within 180 days of baseline
24. Renal failure requiring dialysis or renal transplant
25. Known serious allergy to fluorescein
26. Participation in an investigational study within 30 days prior to baseline that involved treatment with any drug (excluding vitamins and minerals) or device
27. Any women who are pregnant, breast-feeding, or attempting to become pregnant
28. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
BCVA Change | Week 0 to Week 52
  Change in mean BCVA from baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Dilsher S Dhoot, MD, Principal Investigator — California Retina Consultants
Locations (2):
- United States (2):
  - California Retina Consultants - Bakersfield, Bakersfield, California
  - California Retina Consultants - Santa Barbara Office, Santa Barbara, California